CLINICAL TRIAL: NCT01233843
Title: A Phase III Randomized Multicenter Study,Comparing an Induction Chemotherapy Followed by Irradiation and Concurrent Erbitux Versus Chemoradiotherapy for Patients With Locoregional Advanced Head and Neck Cancers
Brief Title: Chemoradiotherapy HNSCC, Randomized Study, Docetaxel,Cisplatin, 5FU,Erbitux.
Acronym: 2007/02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2007-02
Record Dates: First submitted 2010-10-25; First posted 2010-11-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Squamous Cell Head and Neck Carcinoma
Keywords: induction chemotherapy; followed by irradiation and concurrent Erbitux, or radiochemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug and radiation (Other): Radiotherapy : 70 grays , fractionization : 2Gy/day, 5 days / week, for 7 weeks . Concurrent administration of Carboplatin: 70 mg/m2/day (day 1 until day 4)and 5FU 600 mg/m2/day (day 1 until day 4). Weeks 1; 4; 7.
  Interventions: Drug: carboplatin; Drug: 5 fluorouracil; Radiation: radiation therapy
- drug and radiation (Experimental): Induction chemotherapy by Docetaxel 100mg/m2, day 1; cisplatin 100mg/m2, day 1; 5-Fluorouracil 1000mg/m2 (from day 1 to day 5), for a total of three cycles .Those cycles are administrated at day 1; day 22, day43.
  This induction chemotherapy is followed ( for responders or stable disease patients)by radiotherapy (70 grays for 7 weeks) and concurrent Erbitux( weekly administration).
  Interventions: Drug: carboplatin; Drug: 5 fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — 70 mg per m2 and per day for four days. day 1; day 22; day 43
Drug: 5 fluorouracil — 600mg per m2 per day for four days. 3 cycles day 1; day 22; day 43
Radiation: radiation therapy — total dose: 70 grays. The patient receives 2 grays per day; five days a week during 7 weeks

SUMMARY:
The purpose of this study is to demonstrate that induction chemotherapy followed by radiation therapy plus Cetuximab will give better results than the validated treatment (chemoradiotherapy), for treatment of locoregional advanced head and neck cancers.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy (radiotherapy+ carboplatin + 5FU) is a validated treatment for patients with locoregional advanced head and neck cancers.

This study evaluates the outcome of induction chemotherapy (docetaxel, cisplatin, 5 FU) followed by radiation therapy + Erbitux for patients with head and neck carcinoma with almost one measurable lesion by RMI or CT scan.

We hope we can improve the progression free survival of 14% at two years .

ELIGIBILITY:
Inclusion Criteria:

* head and neck locally advanced,non metastatic carcinoma
* not suitable for surgery

Exclusion Criteria:

* non squamous cell head and neck cancer
* previous malignancy
* previous treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Complete response rate of the treatment | by CT scan or MRI and endoscopy 2 years after the end of treatment
  measure of the tumor

SECONDARY OUTCOMES:
The second focus of this study is to compare Overall survival between the two arms . It is defined as the time from the date of randomization to the date of death from any cause. | Date of death
  Aftercare every six months

CONTACTS AND LOCATIONS:
Overall Officials: Lionnel GEOFFROIS, oncologist, Study Director — Centre Alexis Vautrin NANCY France; Etienne BARDET, oncologist, Principal Investigator — Centre Rene Gauducheau NANTES France; Christian SIRE, oncologist, Principal Investigator — Hopital de Bretagne Sud LORIENT France; Laurent MARTIN, oncologist, Principal Investigator — Centre Guillaume le Conquerant LE HAVRE France; Jean-Marc TOURANI, oncologist, Principal Investigator — CHU POITIERS France; Philippe MAINGON, oncologist, Principal Investigator — Centre Georges Francois Leclerc; Ayman ZAWADI, oncologist, Principal Investigator — CHD de Vendee LA ROCHE SUR YON France; François GUICHARD, oncologist, Principal Investigator — Polyclinique de BORDEAUX NORD France; Anne-Françoise DILLIES, oncologist, Principal Investigator — Centre Jean Perrin CLERMONT FERRAND France; Dominique De RAUCOURT, oncologist, Principal Investigator — Centre François Baclesse CAEN France; Emmanuel BABIN, oncologist, Principal Investigator — Hopital Cote de Nacre CAEN France; Claude TUCHAIS, oncologist, Principal Investigator — Centre Paul Papin ANGERS France; XU SHAN Sun, oncologist, Principal Investigator — Hopital Emile Muller MULHOUSE France; Nicolas MEERT, oncologist, Principal Investigator — Grand Hôpital de Charleroi Belgique; Anne-Rose HENRY, oncologist, Principal Investigator — CHU André Vésale MONTIGNY Belgique; Cedrik LAFOND, oncologist, Principal Investigator — Centre Jean Bernard LE MANS France; Thierry PIGNON, oncologist, Principal Investigator — Centre Saint Louis TOULON France; Ali HASBINI, oncologist, Principal Investigator — Clinique Armoricaine SAINT BRIEUC France; Jean BOURHIS, oncologist, Principal Investigator — Institut Gustave Roussy VILLEJUIF France; Marie SALIOU, oncologist, Principal Investigator — Centre Etienne Dolet SAINT NAZAIRE France; Alexandre COUTTE, oncologist, Principal Investigator — CHU sud AMIENS France
Locations (1):
- GIRARD CALAIS Marie-Helene, Tours, France